CLINICAL TRIAL: NCT03787420
Title: Development and Needs Assessment and Efficiency of Smart Communication System for Patients With ALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 107-3011-F-027-002-
Record Dates: First submitted 2018-10-25; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-10

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional communication system (Active Comparator)
  Interventions: Other: communication system
- intelligent communication system (Experimental)
  Interventions: Other: communication system

INTERVENTIONS:
Other: communication system — We will use the questionnaire "Amyotrophic Lateral Sclerosis Supportive Care Needs ,Amyotrophic Lateral Sclerosis Specific Quality of Life Instrument-Revised, Beck Depression Inventory and Caregiver Burden Scale.

SUMMARY:
This project aims to develop a smart communication system for patients with amyotrophic lateral sclerosis (ALS), especially for stage 3 and stage 4 (late stage). Patients with ALS will be able to communicate with outer environment by means of mental control or eye tracking control, which would increase their life quality. This integrated research project includes experts from different domains and proposes a solution for smart communication system.

DETAILED DESCRIPTION:
A multi-function brain- computer interface (BCI) communication system will be developed by combining a BCI system (subproject 1) and a 3D electro-cap (subproject 3). Then, this system and an eye-controlled device (subject 2) are further integrated to a smart communication system. The outputs of the system are presented with the original voice the ALS patients, which will be achieved by using the voice reconstruction technology (subproject 4) in this project. All the user-interfaces of the BCI and eye tracking systems will be re-deigned by employing human factors engineering to increase the usability of the proposed smart communication system for ALS. Finally, the validity of the system in improving the life quality of ALS will be assessed through clinical study.

ELIGIBILITY:
Part one:

Inclusion Criteria:

* ALS diagnostic criteria (Brooks et al., 2000).Must have the following characteristics:

  1. Degeneration of motor neurons (LMN) by clinical, electrophysiological or neuropathological evidence.
  2. Degeneration of upper motor neurons (UMN) is demonstrated by clinical examination.
  3. According to the medical history or examination, the symptoms or signs gradually disappear in a certain part.

Also, there are no features:

1. Electrophysiological or pathological evidence of other diseases that may explain signs of LMN and/or UMN degradation
2. Neuroimaging evidence of other diseases that may explain the observed clinical electrophysiological signs.

   * Use Mandarin as the main language.
   * Age limits minimum is 20

Exclusion Criteria:

* Concomitant other central nervous disorders that interfere with their cognitive function, such as dementia, severe depression, and psychosis.
* The questionnaire cannot be completed without the assistance of others.

Part two:

Inclusion Criteria:

* ALS diagnostic criteria (Brooks et al., 2000).
* Use Mandarin as the main language.
* Age limits minimum is 20
* In everyday oral communication, people who are consciously difficult.
* Ability to perform equipment wear and system operators.

Exclusion Criteria:

* Concomitant other central nervous disorders that interfere with their cognitive function, such as dementia, severe depression, and psychosis.
* After correction, the visual acuity cannot see the communication board.
* The scalp is sensitive or there is deep brain stimulation, etc. It is not applicable to brain wave measurement.
* -The questionnaire cannot be completed without the assistance of others.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Part 1- Amyotrophic Lateral Sclerosis Supportive Care Needs | 30mins
  To comprehensively assess the perceived supportive care needs of patients with ALS.
Part 2 - Amyotrophic Lateral Sclerosis Specific Quality of Life Instrument-Revisedclinical study | one week
  We try to understand the validity of the system. This measurement can help us know that our system could be beneficial or not on the quality of life in patient with ALS.

SECONDARY OUTCOMES:
Part 2 - Beck Depression Inventoryc | one week
  We try to understand the validity of the system. This measurement can help us know that our system could be beneficial or not on the degree of depression of life in patient with ALS.
Caregiver Burden Scale | one week
  We try to understand the validity of the system. This measurement can help us know that our system could be beneficial or not on the burden in patient's caregiver.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Taipei Veterans General Hospital, Taipei, Taiwan